CLINICAL TRIAL: NCT00228319
Title: Antioxidant Effects on the Outcome of Ovarian Cancer
Brief Title: Treatment of Newly Diagnosed Ovarian Cancer With Antioxidants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jeanne Drisko, MD, CNS, FACN (Other)
Collaborators: Cancer Treatment Research Foundation (Other); University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jeanne Drisko, MD, CNS, FACN, Director Integrative Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7823; G-01-029
Record Dates: First submitted 2005-09-23; First posted 2005-09-28 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Ascorbic Acid; Paclitaxel; Carboplatin; Vitamin A; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care Group (Active Comparator): carboplatin and paclitaxel chemotherapy
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Standar of Care + Ascorbic Acid Group (Experimental): carboplatin and paclitaxel chemotherapy, plus intravenous sodium ascorbate. In addition, participants will take a mix of vitamins including oral ascorbic acid, oral mixed natural carotenoids with vitamin A and oral vitamin E.
  Interventions: Dietary Supplement: Oral Ascorbic Acid; Drug: Paclitaxel; Drug: Carboplatin; Drug: Sodium Ascorbate; Dietary Supplement: Oral Mixed natural Carotenoids with Vitamin A; Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Oral Ascorbic Acid — 4 grams per day for 12 months
  Arms: Standar of Care + Ascorbic Acid Group
Drug: Paclitaxel — Six cycles
  Other Names: Taxol; Onxal
Drug: Carboplatin — Six cycles
  Other Names: Paraplatin
Drug: Sodium Ascorbate — Intravenous infusion at 0.5 gram/min twice weekly over 1-2 hours at a dose to achieve levels of 400 mg/dl for 12 months
  Other Names: Vitamin C
  Arms: Standar of Care + Ascorbic Acid Group
Dietary Supplement: Oral Mixed natural Carotenoids with Vitamin A — Capsule containing mixed carotenoids and vitamin A. Participant to take 1 daily for 12 months
  Arms: Standar of Care + Ascorbic Acid Group
Dietary Supplement: Vitamin E — 500 IU per capsule and participant to take 1 capsule daily for 12 months
  Arms: Standar of Care + Ascorbic Acid Group

SUMMARY:
The purpose of this study is to try and understand if there is added benefit or increased harm when antioxidant nutritional supplements are added to traditional chemotherapy in the treatment of ovarian cancer.

DETAILED DESCRIPTION:
The subjects are randomized to 2 study groups. Group 1 receives standard chemotherapy prescribed by the cancer doctor (carboplatin and paclitaxel)with a possible choice to extend chemotherapy for up to an additional 12 months.

Group 2 receives standard chemotherapy in the same manner as group 1. In addition, they receive 12 months of oral or IV nutritional supplements.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed carcinoma of the ovary stage III or IV
* measurable or assessable disease
* drug refractory ovarian cancer
* must be 18 years of age or must have parental consent to enroll in the study
* must be ambulatory

Exclusion Criteria:

* evidence of significant psychiatric disorder by history or exam
* consumption of excess alcohol (more than 4 of any of the following per day: 30 ml distilled spirits, 340 ml beer, or 120 ml wine) or recreational drugs
* tobacco use
* prior treatment with an investigational drug, chemo, radiation therapy, or hormonal therapy within the preceeding month
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Adverse events by NCI CTC version 3.0 | At each oncology clinic visit

SECONDARY OUTCOMES:
Quality of Life Questionnaire | once a month for 6 months and the end of the study
Blood chemistry | At each oncology clinic visit
CA-125 analysis | At each oncology clinic visit
complete CBC with differential | At each oncology clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne A. Drisko, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Result] Ma Y, Chapman J, Levine M, Polireddy K, Drisko J, Chen Q. High-dose parenteral ascorbate enhanced chemosensitivity of ovarian cancer and reduced toxicity of chemotherapy. Sci Transl Med. 2014 Feb 5;6(222):222ra18. doi: 10.1126/scitranslmed.3007154. PMID 24500406